CLINICAL TRIAL: NCT02593214
Title: A Clinical Trial to Asses the Performance and Safety of an Innovative Female Condom (Wondaleaf®) Among Healthy Married Couples
Brief Title: Performance and Safety Trial of an Innovative Female Condom (Wondaleaf®)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Twin Catalyst Sdn. Bhd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NMRR-15-333-24953
Record Dates: First submitted 2015-10-27; First posted 2015-11-02 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2016-08

CONDITIONS: Pregnancy; Sexually Transmitted Disease
Keywords: Condoms, Female; Contraception, Barrier
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wondaleaf Arm (Experimental): This is a single arm clinical trial, all subjects and their married couples were be recruited to the arm using investigational device Wondaleaf only.
  Interventions: Device: Wondaleaf®

INTERVENTIONS:
Device: Wondaleaf® — Use of Wondaleaf® during sexual intercourse with husband for 5 times in a month period

SUMMARY:
General objective:

To assess the performance and safety profile of a novel innovative design of female condom (Wondaleaf®) among healthy married women.

Specific objectives :

* To determine the failure rate of Wondaleaf®, in terms of clinical breakage, non-clinical breakage, invagination, misdirection, and slippage.
* To determine the acceptability and satisfaction of use of Wondaleaf® by subjects and their spouses.
* To assess the safety profile of Wondaleaf®.

DETAILED DESCRIPTION:
This is a single-centre clinical trial to assess the performance and safety profile of Wondaleaf® in healthy married women. Referrals from doctors and nurses in the Maternal and Child Health Clinics, Family Planning Clinics and private clinics in Sibu will be received. A total of 63 couples will be recruited to use Wondaleaf® and to study self-reported total clinical failure and total female condom failure and their components failure events of clinical breakage, non-clinical breakage, total breakage, slippage, misdirection, and invagination (as per World Health Organisation (WHO) Female Condom Technical Review Committee definition(1)). Secondary outcomes were safety parameters (retention of investigational device intra-vaginally should it break, complaint of sexually transmitted diseases, vaginal infection and/or urinary tract infections, all adverse events, serious adverse events, adverse device events and serious adverse device events, allergic reaction) as well as acceptability and satisfaction of the use of Wondaleaf®.

A focus group discussion will be held for the first two couples, to a maximum of five couples recruited based on the same inclusion and exclusion criteria will be asked to trial the process of training / counselling of using the condom, as well as completing the coital log. Experience gathered from these focus group testing and discussion, will be used to enhance the strength of this protocol.

Subsequently, each couple will be asked to use five Wondaleaf® and to complete a coital log at home after each condom use. Before putting on the investigational device, the subject must check for device or package breakage. During sexual intercourse, the couple ought to notice if any breakage of the condom has occurred, and if the female condom slips completely out of the vagina or the penis of male spouse is inserted between the condom and the vaginal wall as well as event of invagination (when the external retention feature of the female condom is partly or fully pushed into the vagina).

Each subject must maintain the wearing of investigational device for the entire process of intercourse until the male spouse ejaculate intra-vaginally. Following each ejaculation of the male spouse, the investigational devices must be checked for breakage before, during and after withdrawal of the condom from the vagina. A coital log must be completed by the couples within 12 hours after the use of each investigational device. Coital logs are used to obtain data for condom performance and safety. The five female investigational devices should be used within a period of four weeks. The used investigational devices shall be discarded safely in the usual and safe manner at home.

After the women completed five uses of Wondaleaf® or after four weeks (whichever occurs first), they will return to the clinic to return their coital log and to fill out an acceptability and satisfaction questionnaire. Any unused female investigational devices (i.e. the female condom) will be returned for counting purposes.

If the women were confirmed pregnant during study period, the subjects will be withdrawn from the study. The married couple will be referred for antenatal care of their choice.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active and legally married couples both between 21 and 45 years of age, and who have been in sexual relationship for at least 6 months;
* Married couples who are willing to participate (i.e. maintain sexually active and agree to have penile-vaginal intercourse with frequency sufficient to meet protocol requirements) and having signed informed consent form;
* Married women willing to have physical examination of the genitalia by the investigator (who is a medical doctor);
* Married women who are willing to take urine pregnancy test;
* Married couples who are planning to get pregnant, but do not mind delaying it;
* Married couples who are not planning for pregnancy soon, yet do not mind getting pregnant (however if found pregnant during the study period, study for the couple will be terminated);
* Married woman and/or her spouse who are on effective contraception (e.g. oral contraceptive, intrauterine device, injectable, patch), or female / male sterilisation methods before entering the study and able to maintain the contraception throughout the study period;
* Married couples who agree to use only study female condom during the time of participation;
* Married couples who are able to understand instructions for correct use of study female condoms;
* Married couples who agree not to use male condom when using the study female condom in a single sexual intercourse;
* Married couples who agree not to use drugs or non-study devices that affect sexual performance;
* Married couples who agree not to wear any genital piercing jewellery while using study female condoms;
* Literate married couple who can complete the study questionnaire and coital log on their own in language of their choice (English, Chinese, or Malay);
* Married couples who are able to comply with completing questionnaire and coital log, as well as attending all study visits.

Exclusion Criteria:

* Female subject with known history of untreated or suspected sexually transmitted infection(s) including HIV/AIDS, vaginal or uterine infection(s), and/or urinary tract infections;
* Female subject with a history of abnormal Pap smear or cervical / uterine diseases;
* Female subject who is pregnant (established by urine pregnancy test), or desires to become so while participating in study;
* Either one of the married couple who have known history of allergy to the devices or materials used to manufacture the investigational devices, or any female or male condom, or lubricants that are used on the devices;
* Those staff who work directly under the investigators and/or employed directly by the device manufacturers, sponsor and study team;
* Female subject who have menopausal symptom (12 months history with no bleeding unless because of contraceptive methods);
* Male subject who has known erectile or ejaculatory dysfunction;
* Either one of the married couple who had history of hospitalisation because of acute illness within three months before Visit 1;
* Either one of the married couple is using any medications or preparation applied topically or intravaginal to the genitalia, other than that supplied for the study (subjects can be rescreened 14 days after the recovery, if the application are for acute illness);
* Any married couple who have received advice from their medical doctor for not engaging in sexual intercourse during the intended study period because of their health conditions, which may include chronic disease or chronic administration (defined as more than 14 days in total) of any medicine, based on medical history and physical examination (no laboratory testing required);
* Women subject and/or their spouse taking medicine which is known to influence sexual performance / libido, or to cause impotence, for any reasons, 30 days before visit 1, and during the intended study period (no laboratory testing required);
* Acute disease at the time of enrolment. Acute disease is defined as the presence of a moderate or severe illness with or without fever. Fever is defined as axillary / tympanic / rectal temperature ≥ 38°C. Subjects can be rescreened 14 days after the recovery;
* Active untreated tuberculosis or communicable diseases of the women subjects and/or their spouse based on medical history;
* Blood dyscrasias, bleeding disorder, leukaemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems;

  . The couple concurrently participating in another clinical study involving female and/or male condom;
* Presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, hepatic, immunologic, hematological, endocrine, or nervous system(s) or psychiatric disease or other conditions that may interfere with the health conditions (such as in case the women subject become pregnant), or would place the subjects at increased risk, as determined by the investigator(s).

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Total female condom failure | Five uses of investigational devices, an average of one month
  Number of times a non-clinical breakage, clinical breakage, or slippage occurs, or that is associated with misdirection, invagination, or any additional failure modes identified in the risk assessment

SECONDARY OUTCOMES:
Total clinical failure | Five uses of investigational devices, an average of one month
  the numbers of female condoms that clinically break or slip, or that are associated with misdirection, invagination, or any additional failure modes identified in the risk assessment, which result in reduction of the protective function of the condom.
Clinical breakage | Five uses of investigational devices, an average of one month
  The number of times a breakage of the condom during sexual intercourse or during withdrawal of the female condom from the vagina (potential adverse clinical consequences) occurs
Non-clinical breakage | Five uses of investigational devices, an average of one month
  Number of times a breakage is noticed before intercourse or occurring after withdrawal of the condom from the vagina (no potential adverse clinical consequences)
Total breakage | Five uses of investigational devices, an average of one month
  the number of all condom breakages at any time before, during, or after sexual intercourse; includes both clinical and non-clinical breakages
Slippage | Five uses of investigational devices, an average of one month
  Number of times when a female condom slips completely out of the vagina during sexual intercourse
Misdirection | Five uses of investigational devices, an average of one month
  Number of times a vaginal penetration whereby the penis is inserted between the condom and the vaginal wall occurs
Invagination | Five uses of investigational devices, an average of one month
  Number of times when the external retention feature of the female condom is partly or fully pushed into the vagina during sexual intercourse
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Five uses of investigational device, an average of one month
  Monitoring of adverse event (locally at the perineum and/or vagina, per vaginal discharge, or any systemic reaction; and local reaction of the penis of the spouse) and adverse device event, as well as if Wondaleaf® ever breaks, if any portion of it retain intra-vaginally
Satisfaction | Five uses of investigational device, an average of one month
  Satisfaction as assessed by the Satisfaction Questionnaire (Beksinska et al, 2013) - which assess using Likert scale ease of condom use/remove, comfort during sex, satisfaction with feeling of sex, in comparison to male condom and no condom, and preference with regards to male condom
Acceptability | Five uses of investigational device, an average of one month
  Acceptability as assessed by four study-designed questions about Wondaleaf on whether Wondaleaf is a useful device for use worldwide and in Malaysia (very useful, moderately useful, not useful); if it is generally acceptable as female condom worldwide and in Malaysia (very acceptable, acceptable, unsure, not acceptable, highly unacceptable).

CONTACTS AND LOCATIONS:
Overall Officials: Teck-Hock Toh, Principal Investigator — Clinical Research Centre, Sibu Hospital, Sarawak State Health Department, Ministry of Health Malaysia; Loke-Meng Ong, Principal Investigator — Clinical Research Centre, Penang General Hospital, Penang State Health Department, Ministry of Health Malaysia; Shirin Hui Tan, Principal Investigator — Clinical Research Centre, Sibu Hospital, Sarawak State Health Department, Ministry of Health Malaysia; Sing Hong Chuo, Principal Investigator — Clinical Research Centre, Sibu Hospital, Sarawak State Health Department, Ministry of Health Malaysia
Locations (1):
- Sibu Hospital, Sibu, Sarawak, Malaysia

REFERENCES:
- [Background] Beksinska M, Joanis C, Manning J, Smit J, Callahan M, Deperthes B, Usher-Patel M. Standardized definitions of failure modes for female condoms. Contraception. 2007 Apr;75(4):251-5. doi: 10.1016/j.contraception.2006.10.003. Epub 2007 Feb 7. PMID 17362701
- [Background] Mitchell HS, Stephens E. Contraception choice for HIV positive women. Sex Transm Infect. 2004 Jun;80(3):167-73. doi: 10.1136/sti.2003.008441. PMID 15169996
- See also: Reproductive Health Supplies Coalition. Caucus on new and underused reproductive health technologies 2013. — http://www.rhsupplies.org/fileadmin/uploads/rhsc/Working_Groups/New_Underused_RH_Technologies_Caucus/Documents/Technical_Briefs/rhsc-brief-female-condom_A4.pdf